CLINICAL TRIAL: NCT03889535
Title: A Comparison of Anterior Pediatric Zirconia Crowns and Bonded Composite Resin Strip Crowns: A One-year Feasibility Study
Brief Title: Anterior Zirconia vs. Resin Strip Crowns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Michael Casas, Dentist-in-Chief, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1000062660
Record Dates: First submitted 2019-03-21; First posted 2019-03-26 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Caries, Dental
Keywords: primary maxillary incisors; crowns; bonded composite resin strip crowns; zirconia crowns; one-year survival
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resin strip crowns (Active Comparator): Current standard full coverage restoration provided for primary incisors. Please see intervention section for detailed description of technique.
  Interventions: Device: Resin strip crowns
- Zirconia crowns (Experimental): Experimental treatment under study. Zirconia crowns are an alternative restorative option. Please see intervention section for detailed description of technique.
  Interventions: Device: Zirconia crowns

INTERVENTIONS:
Device: Resin strip crowns — Technique:
  I.Select shade of resin-based composite II.Rubber dam isolation III.Select primary incisor celluloid crown form with mesiodistal width similar to the tooth to be restored and trim the selected crown form to fit.
  IV.Remove decay with slow speed round bur. Perform pulp therapy, if indicated. V.Reduce incisal edge by 1.5 mm VI.Reduce interproximal surfaces by 0.5 to 1.0 mm with feather edge at gingival margin. The interproximal walls should be approximately parallel.
  VII.Reduce buccal surface by 1.0 mm and lingual surface by 0.5 mm with feather edge at gingival margins.
  VIII. Round line angles IX.Etch for 15 to 20 seconds, rinse and air dry X. Apply bond and polymerise XI. Fill crown form to 2/3 full with composite resin and seat onto the tooth. Remove excess material with hand instrument. Polymerise.
  XII. Remove celluloid crown form with scaler XIII. Finish and polish
  Arms: Resin strip crowns
Device: Zirconia crowns — I.Choose appropriately sized crown based on tooth's dimension; evaluate occlusion. II.Rubber dam isolation. III.Remove decay, perform pulp therapy if indicated. IV.Prep mesial half of incisal edge to complete thickness of 001 donut bur. V.Prep and blend distal half of incisal edge to create uniform incisal reduction. VI. Create chamfer margin at gum line at least half the thickness of bur tip. VII. Taper incisal half lingually to create a thin incisal edge. VIII. Remove cingulum and 0.75-1.25mm of lingual enamel; blend together forming smooth, slightly concave surface extending to tissue. IX. Thin incisal half. X.With 004 flame bur, remove chamfer margin at tissue level. Keep bur parallel to long axis of tooth. Remove chamfer in incremental steps, XI. Extend tip of bur full 2mm subgingivally. While hugging bur axially along root surface, make 3 circumferential passes. XII.Clean tooth and control bleeding. XIII.Cement crown with pure glass ionomer cement
  Arms: Zirconia crowns

SUMMARY:
This study is comparing the effectiveness of two different dental crown fillings (resin crowns and zirconia crowns) for primary front teeth (incisors). Both dental crown fillings are currently used by community pediatric dentists. Resin crowns are currently the standard treatment for primary incisors at The Hospital for Sick Children (SickKids). Zirconia crowns are not presently used at SickKids. It is unknown if one type of crown is better than the other type. If the zirconia crowns produce similar or better results in fixing the primary front teeth, then the zirconia crowns may become the new standard of care at SickKids.

DETAILED DESCRIPTION:
To assess the clinical outcome of pediatric zirconia crowns and to provide evidence-based treatment, a prospective, well controlled study would be beneficial. Due to a lack of existing outcome data for bonded resin strip crowns and zirconia crowns, a feasibility study is indicated to establish the basis for randomized controlled trial design. The goal of this feasibility study is to compare the clinical outcomes of the zirconia crowns and bonded composite resin strip crowns in primary maxillary incisors. Therefore the aims of the research study is as follows:

1. To statistically compare the one-year survival of resin composite strip crowns and zirconia crowns in primary maxillary incisors.
2. To statistically compare the frequency of pulp therapy required for placement of zirconia crowns and resin composite strip crowns in primary maxillary incisors.
3. To measure the frequency at which teeth randomized to zirconia crowns are deemed restorable with strip crowns and not zirconia crowns, and vice versa.

After induction of general anesthesia, following the confirmation that incisor(s) can be restored by the treating dentist, each study participant will be randomly allocated to either the strip crown or the zirconia crown group. The assignment will be done using a computer-generated simple random number sequence with a one to one allocation ratio. The treatment will be consistent for each patient for all eligible teeth, although the experimental unit is the incisor.

Each research participant will be reassessed clinically at 6 and 12 months after treatment. Follow-up appointments will be scheduled by the Department of Dentistry at the Hospital for Sick Children (SickKids). Clinical reassessment will be conducted by one investigator. Intra-oral photographs will be acquired at 6 months and at 12 months. All photographs will be taken by the same investigator, using a standardized imaging format. Two photographs per patient will be acquired: one extra-oral photograph, limited to the maxillary right cuspid (tooth 53) to left cuspid (tooth 63); and one extra-oral maxillary occlusal photograph, limited to the maxillary right cuspid (tooth 53) to left cuspid (tooth 63). Photographs will be taken with a Canon Rebel XSi and a Canon ring flash Macro Ring Lite MR-14EX II.

Parents will also take 2 photographs of their child's teeth using their own camera or phone. They will be provided with an example of how to take those photographs. They will send the photographs to the investigators via a secured SickKids e-mail. Only the research investigators and the research coordinator will have access to the secured e-mail. Pictures sent by the parents will be stored on a the photograph and X-ray database at SickKids. A reminder to take the pictures at 6 and 12 months after the surgery will be sent using the secured e-mail. Photographs taken by the parents will be used for the photographic assessment if clinical photographs are unsuccessful at the follow-ups and if they are of sufficient quality for assessment based on the investigators' judgment.

ELIGIBILITY:
Inclusion Criteria:

1. Incisors with large carious lesions not restorable with intra-coronal restorations
2. Incisors that have received pulp therapy
3. Incisors that have been fractured and have lost an appreciable amount of tooth structure
4. Incisors with multiple hypoplastic defects or developmental disturbances
5. Incisors with small interproximal lesions with large areas of cervical decalcification

Exclusion Criteria:

1. Patient is classified as American Society of Anesthesiologists (ASA) III or higher
2. Caries associated with signs and symptoms of irreversible pulpitis and/or clinical evidence of an odontogenic infection
3. There is radiographic evidence of pathological root resorption, root fracture secondary to trauma or periapical radiolucency, iv) lacking adequate dental coronal structure to allow restoration with full coverage restoration
4. Patient has non-English speaking parents.

Ages: 18 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Survival outcome | 12 months
  The survival outcome will consist of clinical assessment and photographic assessment. One investigator will clinically assess the incisors for restoration survival. The assessed criteria are: presence of the tooth (teeth lost prior to general anesthesia or during general anesthesia will be excluded from statistical analysis), presence of the restoration, integrity of the restoration, recurrent decay and discoloration. Two blinded disinterested expert raters (staff pediatric dentists) will assess the photographs for restoration survival.

SECONDARY OUTCOMES:
Frequency of pulp therapy | 1 day (Day of crown restoration)
  On the day of treatment under general anesthesia, the treating dentist, the dental assistant or the nurse will fill out the pulpotomy data collection form. Each treated tooth will be marked as having received a pulpotomy (P), or not having received a pulpotomy (X).
Treatment plan alteration | 1 day (Day of crown restoration)
  On the day of treatment under general anesthesia, the treating dentist, the dental assistant or the nurse will fill out the restorative treatment data collection form. Each form will be filled with the randomly assigned treatment and the completed treatment: zirconia crowns (ZC) or composite resin strip crowns (CRSC). It will be determined if patient received the treatment originally assigned and reason for deviation from randomly selected treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Casas, DDS, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Michael Joseph Casas, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual Patient Data (IPD) will not be shared with other researchers

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT03889535/Prot_SAP_000.pdf